CLINICAL TRIAL: NCT05067595
Title: A Randomized, Controlled, Phase I Study of Fecal Microbiota Transplant and Dietary Fiber Supplementation in Graft Versus Host Disease
Brief Title: Fecal Microbiota Transplant and Dietary Fiber Supplementation for the Treatment of Gut Graft Versus Host Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RG1006202; NCI-2019-07698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10276 (Other: Fred Hutch/University of Washington Cancer Consortium); 1R01HL166107 (NIH)
Record Dates: First submitted 2019-12-10; First posted 2021-10-05 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Intestinal Graft Versus Host Disease
MeSH Terms: interventions — Colonoscopy; Fecal Microbiota Transplantation; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Arm I (upper FMT) (Experimental): Patients receive upper FMT capsules PO over 5 days or via post-pyloric or NG feeding tube over 2 days. Patients also undergo tissue, stool, stool swabs, and blood sample collection throughout the study.
  Interventions: Biological: Fecal Microbiota Transplantation; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm II (Lower FMT) (Experimental): Patients undergo lower FMT via colonoscopy on day 0. Patients also undergo tissue, stool, stool swabs, and blood sample collection throughout the study.
  Interventions: Procedure: Colonoscopy; Biological: Fecal Microbiota Transplantation; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm III (upper FMT, fiber supplementation) (Experimental): Patients receive upper FMT capsules PO over 5 days or via post-pyloric or NG feeding tube over 2 days. Patients also receive fiber supplementation PO or via post-pyloric or NG feeding tube from the first day of FMT administration and up to 6 weeks post FMT. Patients also undergo tissue, stool, stool swabs, and blood sample collection throughout the study.
  Interventions: Biological: Fecal Microbiota Transplantation; Dietary Supplement: Nutritional Supplementation; Other: Survey Administration; Procedure: Biospecimen Collection
- Arm IV (Lower FMT, fiber supplementation) (Experimental): Patients undergo lower FMT via colonoscopy on day 0. Patients also receive fiber supplementation PO or via post-pyloric or NG feeding tube from day 0 up to 6 weeks post FMT. Patients also undergo tissue, stool, stool swabs, and blood sample collection throughout the study.
  Interventions: Procedure: Colonoscopy; Biological: Fecal Microbiota Transplantation; Dietary Supplement: Nutritional Supplementation; Other: Survey Administration; Procedure: Biospecimen Collection

INTERVENTIONS:
Procedure: Colonoscopy — Undergo lower FMT via colonoscopy
  Arms: Arm II (Lower FMT); Arm IV (Lower FMT, fiber supplementation)
Biological: Fecal Microbiota Transplantation — Given upper FMT PO or via post-pyloric or NG feeding tube
  Other Names: Fecal Material Transplantation; Fecal Transplantation; FMT; Poo Transplant; Poop Transplant; Stool Transplant
  Arms: Arm I (upper FMT); Arm III (upper FMT, fiber supplementation)
Biological: Fecal Microbiota Transplantation — Undergo lower FMT via colonoscopy
  Other Names: Fecal Material Transplantation; Fecal Transplantation; FMT; Poo Transplant; Poop Transplant; Stool Transplant
  Arms: Arm II (Lower FMT); Arm IV (Lower FMT, fiber supplementation)
Dietary Supplement: Nutritional Supplementation — Given dietary fiber supplementation PO or via post-pyloric or NG feeding tube
  Other Names: Supplementation
  Arms: Arm III (upper FMT, fiber supplementation); Arm IV (Lower FMT, fiber supplementation)
Other: Survey Administration — Ancillary studies
Procedure: Biospecimen Collection — Undergo tissue, stool, stool swabs, and blood sample collection
  Other Names: Biological Sample Collection

SUMMARY:
This phase I trial studies how well fecal microbiota transplant and dietary fiber supplementation work in treating patients with gut graft versus host disease. Fecal microbiota transplant entails inoculating donor stool into a recipient's gastrointestinal tract. Changing the gut microbiome by fecal microbiota transplant and fiber supplementation may help treat gut graft versus host disease.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 4 arms.

ARM I: Patients receive upper FMT capsules orally (PO) over 5 days or via post-pyloric or nasogastric (NG) feeding tube over 2 days.

ARM II: Patients undergo lower FMT via colonoscopy on day 0.

ARM III: Patients receive upper FMT capsules PO over 5 days or via post-pyloric or NG feeding tube over 2 days. Patients also receive fiber supplementation PO or via post-pyloric or NG feeding tube from the first day of FMT administration and up to 6 weeks post FMT.

ARM IV: Patients undergo lower FMT via colonoscopy on day 0. Patients also receive fiber supplementation PO or via post-pyloric or NG feeding tube from day 0 up to 6 weeks post FMT.

Patients also undergo tissue, stool, stool swabs, and blood sample collection throughout the study.

After completion of study treatment, patients are followed up for 365 days.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* History of allogeneic hematopoietic stem cell transplant in the past 365 days
* Post-engraftment, defined by time period following three consecutive days of sustained neutrophil engraftment with an absolute neutrophil count of at least 500 cells/mm^3
* Mild to severe acute GI GvHD, at least stage 1, as measured by one of the following:

  * Modified Glucksberg criteria for GI GvHD averaged over 3 consecutive days and without another explanation for diarrhea such as laxative use or infection. In patients who have already had GI biopsy, biopsy histology must be compatible with GVHD, although biopsy is not required
  * Biopsy evidence of GI GVHD in the upper or lower GI tract

Exclusion Criteria:

* History of previous serious adverse events associated with FMT
* History of bowel perforation in the last 90 days
* History of gastrointestinal resection in the last 90 days
* History of intestinal obstruction in the last 90 days
* History of diverticulitis in the last 90 days
* History of celiac disease confirmed by serologic testing or small bowel biopsy
* History of severe dietary allergy as designated by World Allergy Organization Subcutaneous Immunotherapy Systemic Reaction Grading System grade 2 or more
* Subjects who are cytomegalovirus (CMV) seronegative at the time of enrollment as indicated by clinical testing unless the fecal microbiota transplant (FMT) donor is CMV seronegative with negative plasma polymerase chain reaction (PCR) assays for CMV.
* Known allergies to loperamide, sodium chloride, glycerol, theobroma oil, hide bovine gelatin, sodium lauryl sulfate, colorants FD&C, titanium dioxide, polyethylene glycol, sodium sulfate, sodium bicarbonate, sodium phosphate, benzalkonium chloride, disodium EDTA or potassium chloride.
* Currently pregnant, planning to become pregnant or breastfeeding during the study period. Women of childbearing potential (those who are not post-menopausal or post-hysterectomy) must be negative for pregnancy per urine pregnancy test at enrollment
* Individuals with the ability to conceive children who are not willing to abstain from sexual activity or use an effective form of birth control during the duration of the study
* Unwilling or unable to participate in study procedures including oral intake of FMT, colonoscopy, fiber supplementation, collection of stool samples and completion study surveys
* Cannot reasonably and safely participate in the study in the opinion of the investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Bacterial composition of stool | At baseline
  Analyses will consist of summary statistics of the bacterial diversity in the microbiome (e.g., the alpha diversity, the abundance of bacterial species associated with protection from graft versus host disease [GvHD]).
Bacterial genes in stool | At baseline
  Specifically abundance of genes related to fiber fermentation and short chain fatty acids production metabolites in stool, specifically short chain fatty acids will be assessed.
Incidence of adverse events | Up to 3 years
  Will by assessed by computing the total number of adverse events (AE)s and serious adverse events (SAE)s, the number per patient, and the number of patients with at least one event. The type of AE/SAE and whether the AE/SAE is related to the fecal microbiota transplant (FMT) or not will be tabulated. These summaries will be computed overall as well as by randomization arm and stratification factor (steroid-responsive, versus steroid-dependent or -refractory disease status). The odds will be compared of at least one SAE per patient by randomization arm and stratification factor using logistic regression with independent variables for route of FMT administration, fiber supplementation, and steroid-responsive, versus steroid-dependent or -refractory disease status. Interaction terms will be considered between these factors and may use exact or firth logistic regression in the event that some categories have zero patients with a SAE.

SECONDARY OUTCOMES:
Complete response (CR) after the initial FMT | At day 28
  Will be defined by stage 0 on the Modified Glucksberg GvHD scale, without abdominal pain or hematochezia. To account for variability in this measure, patient stool volume (inpatients only) and survey data (both inpatients and outpatients) from days 25-27 will be used to determine whether patients meet these criteria or not. Inpatients will be a compare measured stool volumes to those reported via survey, to assess how well the survey data may serve as a surrogate for stool volume. Subjects who die before day 28 will be counted as no CR. The number and proportion of patients with CR by steroid-responsive, versus steroid-dependent or -refractory disease status, and each randomization arm (route of FMT administration and receipt of fiber supplementation) as well as within combinations of these factors will be computed. To test for differences in CR by these factors, logistic regression models similar to those described above for SAE comparisons.
CR or partial response (PR) after the initial FMT | At day 28
  Will be assessed by CR or PR at day 28 will use similar analysis methods as to the CR at day 28 outcome analysis.
Gut and overall GvHD grade | Up to 6 months
  Will be assessed using the Modified Glucksberg scale measurements at baseline and throughout follow-up to summarize decrease in stool volume. For both of these ordinal outcomes (GvHD grade and Modified Glucksberg scale stage), descriptive statistics and graphical summaries to show changes over time by stratification factor and randomization arm. Generalized linear mixed effects models to test for differences in these outcomes by stratification factor and randomization arm.
Six-month survival | At 6 months
  Will be evaluated using Kaplan-Meier curves and Cox proportional hazards regression with independent variables for the steroid- responsive, versus steroid-dependent or - refractory disease and randomization arm as specified in previous models.
Quality of life | Up to 3 years
  Will be summarized at baseline and during study using descriptive statistics.
Decrease in stool volume | Up to 6 months
Levels of MAIT cells in the periphery | Up to 6 months
  Will be assessed using plot cell counts and percentage of lymphocytes for MAIT cells over time to compare longitudinal patterns by study arm and stratification factor. Mann-Whitney tests will be used to evaluate differences in cell counts and percentage of lymphocytes for MAIT cells in recipients of upper versus lower FMT, and individuals who receive fiber supplementation versus those who do not at specific time points post-FMT. Linear mixed effects models may be used to test for differences in longitudinal patterns of these outcomes by randomization arm and stratification factor.
Levels of Treg cells in the periphery | Up to 6 months
  Will be assessed using plot cell counts and percentage of lymphocytes for Treg cells over time to compare longitudinal patterns by study arm and stratification factor. Mann-Whitney tests will be used to evaluate differences in cell counts and percentage of lymphocytes for Tregs in recipients of upper versus lower FMT, and individuals who receive fiber supplementation versus those who do not at specific time points post-FMT. Linear mixed effects models may be used to test for differences in longitudinal patterns of these outcomes by randomization arm and stratification factor.

CONTACTS AND LOCATIONS:
Overall Officials: David Fredricks, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No